CLINICAL TRIAL: NCT00797251
Title: A Novel Simple Technique for Performing Anatomical Right Posterior Sectionectomy of the Liver: the Ultrasound-Guided Finger Compression
Brief Title: Anatomical Right Posterior Sectionectomy of the Liver by IOUS-Guided Finger Compression
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Milan (Other)
Responsible Party: Guido Torzilli, MD, PhD, University of Milan School of Medicine
Other Study IDs: IOUS-Compression
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Colorectal Liver Metastases; Hepatocellular Carcinoma; Liver Malignancies
Keywords: Colorectal liver metastasis; hepatocellular carcinoma; liver surgery; intraoperative ultrasound; finger-compression
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Right posterior section group: Patients with tumors in the right posterior section of the liver (segments 6-7)
  Interventions: Procedure: Anatomical right posterior sectionectomy of the liver by IOUS-guided finger compression.

INTERVENTIONS:
Procedure: Anatomical right posterior sectionectomy of the liver by IOUS-guided finger compression. — The technique consists in IOUS-guided finger compression of the right posterior portal pedicle at the level closest to the tumor but oncologically suitable. This method allows us to anatomically mark the area of resection with nor hilar plate nor IOUS-guided puncture of vessels, which are up to date the only two techniques available to perform anatomical right posterior sectionectomy - namely the removal of segment 6 and 7.
  Other Names: anatomic resection of segment 6-7

SUMMARY:
The use of intraoperative ultrasound (IOUS) allows us to perform new conservative hepatectomies. The investigators previously reported the systematic subsegmentectomy by IOUS-guided finger compression for segments 2-3, which is currently applied for patients with hepatocellular carcinoma (HCC)on cirrhosis. The investigators herein describe a novel technique, which consists in the systematic right posterior sectionectomy by IOUS-guided finger compression.

DETAILED DESCRIPTION:
A novel technique for the demarcation of the resection area by means of IOUS-guided finger compression to accomplish a right posterior sectionectomy is described. Dissection or encirclement of the sectional pedicles for resection area demarcation is thus avoided. Ten patients underwent this technique successfully without mortality or major morbidity. IOUS-guided finger compression of sectional portal pedicle feeding the right posterior section is a feasible, safe, and effective method.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tumors at least at 1 cm distally to the bifurcation of the right portal vein (bifurcation of P5-8 and P6-7) eligible for right posterior sectionectomy, namely the anatomical removal of segment 6 and 7, were considered potential candidates to this procedure. Precisely, these criteria were adopted:

  * Patients with hepatocellular carcinoma (HCC) with infiltrative growing pattern in contact with P6-7;
  * Patients with any type of HCC in contact with P6-7 with distal bile duct dilation;
  * Patients with colorectal liver metastasis (CLM) in contact with P6-7.

Exclusion Criteria:

* Exclusion criteria for carrying out the herein described procedure was considered the presence of tumoral thrombosis in P6-7.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population include patients with primary or secondary liver tumors in the right posterior section of the liver eligible to a right posterior sectionectomy as a primary surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the safety of the anatomical right posterior sectionectomy performed IOUS-guided finger compression. | 6 months

SECONDARY OUTCOMES:
The secondary outcome is the efficacy of the anatomical right posterior sectionectomy performed by IOUS-guided finger compression. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — University of Milan School of Medicine, IRCCS Istituto Clinico Humanitas
Locations (1):
- University of Milan School of Medicine, IRCCS Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Torzilli G, Donadon M, Marconi M, Botea F, Palmisano A, Del Fabbro D, Procopio F, Montorsi M. Systematic extended right posterior sectionectomy: a safe and effective alternative to right hepatectomy. Ann Surg. 2008 Apr;247(4):603-11. doi: 10.1097/SLA.0b013e31816387d7. PMID 18362622
- [Background] Torzilli G, Donadon M, Montorsi M. The surgical margin in liver resection for hepatocellular carcinoma: a real problem or not? Ann Surg. 2007 Oct;246(4):690-1; author reply 691-2. doi: 10.1097/SLA.0b013e318156e286. No abstract available. PMID 17893508
- [Background] Torzilli G, Montorsi M, Del Fabbro D, Palmisano A, Donadon M, Makuuchi M. Ultrasonographically guided surgical approach to liver tumours involving the hepatic veins close to the caval confluence. Br J Surg. 2006 Oct;93(10):1238-46. doi: 10.1002/bjs.5321. PMID 16953487
- [Background] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Background] Torzilli G, Makuuchi M. Ultrasound-guided finger compression in liver subsegmentectomy for hepatocellular carcinoma. Surg Endosc. 2004 Jan;18(1):136-9. doi: 10.1007/s00464-003-9024-x. Epub 2003 Nov 21. PMID 14625736
- [Background] Takasaki K, Kobayashi S, Tanaka S, Saito A, Yamamoto M, Hanyu F. Highly anatomically systematized hepatic resection with Glissonean sheath code transection at the hepatic hilus. Int Surg. 1990 Apr-Jun;75(2):73-7. PMID 2166006
- [Background] Launois B, Jamieson GG. The posterior intrahepatic approach for hepatectomy or removal of segments of the liver. Surg Gynecol Obstet. 1992 Feb;174(2):155-8. PMID 1734576
- [Background] Makuuchi M, Hasegawa H, Yamazaki S. Ultrasonically guided subsegmentectomy. Surg Gynecol Obstet. 1985 Oct;161(4):346-50. PMID 2996162